CLINICAL TRIAL: NCT05697627
Title: Cognitive Training Video Game to Target Subclinical Depressive Symptoms in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hannah Becker, MS, Doctoral Candidate in Clinical Science, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00227345
Record Dates: First submitted 2023-01-07; First posted 2023-01-26 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Depression; Subclinical Depressive Symptoms
Keywords: Cognitive Training Video Game
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Computerized cognitive training (CCT) using EndeavorRx (Experimental): Exciting, youth-friendly computer game, EndeavorRx engages and trains cognitive control across component processes of attention, response inhibition, shifting and working memory.
  Interventions: Device: Computerized cognitive training (CCT) using EndeavorRx

INTERVENTIONS:
Device: Computerized cognitive training (CCT) using EndeavorRx — The EndeavorRx video game is a digital therapeutic designed to improve attention and related cognitive control processes by training interference management.
  ~25 minutes of EndeavorRx video game play per day, for 5 days/week, for up to 4 weeks

SUMMARY:
The purpose of the study is to determine how cognitive control training (CCT) changes behavior in youth with subclinical depressive symptoms. This research will show what types of behavior changes are important for CCT to help reduce depressive symptoms. In the future, this information will be used to try to improve prevention of the development of depression, so that it can help more patients.

DETAILED DESCRIPTION:
The primary study investigator acknowledges contributions from Kate Fitzgerald, Emily Bilek, Christopher Monk, and Adriene Beltz.

ELIGIBILITY:
Inclusion criteria:

1. Parent or guardian willing to give informed consent, and children willing to give informed assent to participate in the study.
2. Males and females (age 9 - 17.99)
3. Participant is willing to engage in a technology-based intervention (technology will be provided to participants who live in the state of Michigan, if not already accessible to participant).
4. Self-reported depressive symptoms (Children's Depression Inventory [CDI] score between 3-19 at Assessment 1)
5. Participants will be required to maintain a stable dose of medications

EXCLUSION CRITERIA

1. Color blindness
2. Unable to play the video game for any reason
3. Current Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) diagnosis of clinical depression, psychosis, or Autism Spectrum Disorder
4. Has enrolled in new psychotherapy (for the treatment of a mood or anxiety disorder) or had changes to their psychotherapy in the 4-weeks prior to study enrollment
5. Endorses items #1, #2, #3, #4, #5, or #6 on the Columbia Suicide Severity Rating Scale (C-SSRS) Screener (Past-Month); i.e., has present suicidal intention/behavior.
6. Has had any changes to their medication in the 4-weeks prior to study enrollment

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Becker, M.S., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
contact

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 participants signed consent forms. During the pre-assignment phase of the study, participants completed several diagnostic and clinical assessments to see if they met eligibility criteria. 11 of these 31 individuals were not assigned to the intervention because of the following: did not meet eligibility criteria (n=9); lost to follow-up during pre-assignment (n=1); the study concluded prior to the assignment phase for this individual (n=1).
Groups:
- Computerized Cognitive Training (CCT) Using EndeavorRx: The EndeavorRx video game is a digital therapeutic designed to improve attention and related cognitive control processes by training interference management. Participants engage in approximately ~25 minutes of EndeavorRx video game play per day, for 5 days/week, for up to 4 weeks.
Period: Overall Study
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Computerized Cognitive Training (CCT) Using EndeavorRx: The EndeavorRx video game is a digital therapeutic designed to improve attention and related cognitive control processes by training interference management. Participants were instructed to engage in approximately 25 minutes of EndeavorRx video game play per day, for 5 days/week, for up to 4 weeks.
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms as Measured by Children's Depression Inventory (CDI)
Description: The CDI was a self-report, 27 item scale used to measure depressive symptoms. Total scores on the CDI ranged from 0 (no depressive symptoms) to 54 (extremely severe depressive symptoms). Higher scores indicated worse depressive symptoms. CDI scores were collected from participants at three timepoints: 1) baseline, 2) approximately 5 weeks after baseline, and 3) up to 4 months after baseline. Results reflect CDI scores collected at the first and second timepoints.
Time Frame: Baseline and approximately 5 weeks after
Population: One participant dropped out of the study before the follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 20
score on a scale
  Baseline CDI scores | 8.85 (3.65)
  Approximately 5 weeks: number analyzed (Participants) | 19
  Approximately 5 weeks | 5.84 (4.37)

2. Primary Outcome: Change in Depressive Symptoms as Measured by Children's Depression Rating Scale - Revised (CDRS-R)
Description: The CDRS-R is a clinician-administered tool used to assess the severity of depression in children and adolescents based on a 17-item scale of depressive symptoms. Total raw scores on this scale range from 17-113, with 17 indicating no or minimal depressive symptoms and 113 indicating extremely severe symptoms of depression. CDRS-R scores were collected from participants at three timepoints: 1) baseline, 2) approximately 5 weeks after baseline, and 3) up to 4 months after baseline. Results reflect CDRS-R scores collected at the first and second timepoints.
Time Frame: Baseline and approximately 5 weeks after
Population: One participant dropped out of the study before the 5-week assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 20
score on a scale
  Baseline - Raw CDRS-R scores | 30.00 (5.69)
  Approximately 5 weeks - Raw CDRS-R scores: number analyzed (Participants) | 19
  Approximately 5 weeks - Raw CDRS-R scores | 24.05 (3.29)

3. Primary Outcome: Change in Cognitive Control Capacity - Overall Reaction Time (RT) Stroop
Description: The Stroop task assesses cognitive control and emotion regulation over emotional information processing by measuring how quickly individuals name the ink color of words that are emotionally-charged or neutral. For this measure, lower scores indicated better performance, i.e., better cognitive control and emotion regulation. Results reflect the average reaction time across all trials of the Stroop task that participants completed.
Time Frame: Baseline and approximately 5 weeks after
Population: 1 person did not complete the baseline cognitive assessment and also withdrew prior to follow-up assessment.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Computerized Cognitive Training (CCT) Using EndeavorRx: Exciting, youth-friendly computer game, EndeavorRx engages and trains cognitive control across component processes of attention, response inhibition, shifting and working memory.
  Computerized cognitive training (CCT) using EndeavorRx: The EndeavorRx video game is a digital therapeutic designed to improve attention and related cognitive control processes by training interference management.
  ~25 minutes of EndeavorRx video game play per day, for 5 days/week, for up to 4 weeks
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 19
milliseconds
  Overall RT on Stroop Task pre-intervention | 1019.44 (131.07)
  Overall RT on Stroop Task post-intervention | 1018.28 (140.31)

4. Primary Outcome: Change in Cognitive Control Capacity - Conflict RT Stroop
Description: The Stroop task assesses cognitive control and emotion regulation over emotional information processing by measuring how quickly individuals name the ink color of words that are emotionally-charged or neutral. For this measure, lower scores indicated better performance, i.e., better cognitive control and emotion regulation. Results reflect the difference in the reaction time between incongruent trials and congruent trials on the Stroop task.
Time Frame: Baseline and approximately 5 weeks after
Population: 1 person did not complete the baseline cognitive assessment and also withdrew prior to follow-up assessment.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 19
milliseconds
  Conflict RT (Incongruent Trial RT - Congruent Trial RT) on Stroop Task pre-intervention | 65.95 (58.60)
  Conflict RT (Incongruent Trial RT - Congruent Trial RT) on Stroop Task post-intervention | 62.32 (96.70)

5. Primary Outcome: Change in Cognitive Control Capacity - Overall RT Flanker
Description: The Flanker task is a psychological experiment that assesses a person's ability to focus on a target stimulus while ignoring distracting stimuli. For this measure, higher scores indicate better performance. Results reflect the average reaction time across all trials of the Flanker task that participants completed at this timepoint.
Time Frame: Baseline and approximately 5 weeks after
Population: Only 19 participants completed any of the cognitive tasks at baseline or follow up. From the 19, 2 participants at pre-intervention did not complete the Flanker task. From the 19, 1 participant at post-intervention did not complete the Flanker task.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 18
milliseconds
  Overall RT on Flanker Task pre-intervention: number analyzed (Participants) | 17
  Overall RT on Flanker Task pre-intervention | 785.93 (266.25)
  Overall RT on Flanker Task post-intervention | 778.62 (435.33)

6. Primary Outcome: Change in Cognitive Control Capacity - Conflict RT Flanker
Description: The Flanker task is a psychological experiment that assesses a person's ability to focus on a target stimulus while ignoring distracting stimuli. For this measure, higher scores indicate better performance. Results reflect the difference in the reaction time between incongruent trials and congruent trials of the Flanker task.
Time Frame: Baseline and approximately 5 weeks after
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 18
milliseconds
  Conflict RT (Incongruent Trial RT - Congruent Trial RT) on Flanker Task pre-intervention: number analyzed (Participants) | 17
  Conflict RT (Incongruent Trial RT - Congruent Trial RT) on Flanker Task pre-intervention | 151.31 (188.11)
  Conflict RT (Incongruent Trial RT - Congruent Trial RT) on Flanker Task post-intervention | 311.82 (970.06)

7. Secondary Outcome: Children's Depression Inventory (CDI) at Third Timepoint
Description: The CDI was a self-report, 27 item scale used to measure depressive symptoms. Total scores on the CDI ranged from 0 (no depressive symptoms) to 54 (extremely severe depressive symptoms). Higher scores indicated worse depressive symptoms. CDI scores were collected from participants at three timepoints: 1) baseline, 2) approximately 5 weeks after baseline, and 3) up to 4 months after baseline. Results reflect CDI scores collected at the third timepoint.
Time Frame: Up to 4 months
Population: The third timepoint was offered as optional to participants and then eventually removed from the protocol altogether. 10 participants returned and completed the CDI at the optional third time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 10
score on a scale | 6.30 (6.48)

8. Secondary Outcome: Depressive Symptoms as Measured by Children's Depression Rating Scale - Revised (CDRS-R) at Third Timepoint
Description: The CDRS-R is a clinician-administered tool used to assess the severity of depression in children and adolescents based on a 17-item scale of depressive symptoms. Total raw scores on this scale range from 17-113, with 17 indicating no or minimal depressive symptoms and 113 indicating extremely severe symptoms of depression. CDRS-R scores were collected from participants at three timepoints: 1) baseline, 2) approximately 5 weeks after baseline, and 3) up to 4 months after baseline. Results reflect CDRS-R scores collected at the third timepoint.
Time Frame: Up to 4 months
Population: The third timepoint was offered as optional to participants and then eventually removed from the protocol altogether. 11 participants returned to complete the CDRS-R for the optional third timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 11
score on a scale | 23.27 (3.82)

9. Secondary Outcome: Cognitive Control Capacity - Overall Reaction Time (RT) Stroop
Description: The Stroop task assesses cognitive control and emotion regulation over emotional information processing by measuring how quickly individuals name the ink color of words that are emotionally-charged or neutral. For this measure, lower scores indicated better performance, i.e., better cognitive control and emotion regulation. Results reflect the average reaction time across all trials of the Stroop task that participants completed at this timepoint.
Time Frame: Up to 4 months
Population: The third timepoint was offered as optional to participants and then eventually removed from the protocol altogether. 11 participants completed the third timepoint assessment, and 6 participants completed the cognitive tasks at this timepoint (including Stroop).
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 6
milliseconds | 982.60 (70.39)

10. Secondary Outcome: Cognitive Control Capacity - Conflict RT Stroop
Description: as for outcome 4
Time Frame: Up to 4 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 6
milliseconds | 58.45 (76.85)

11. Secondary Outcome: Cognitive Control Capacity - Overall RT Flanker
Description: as for outcome 5
Time Frame: Up to 4 months
Population: The third timepoint was offered as optional to participants and then eventually removed from the protocol altogether. 11 participants completed the third timepoint assessment, and 6 participants completed the cognitive tasks at this timepoint (including Flanker).
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 6
milliseconds | 597.31 (93.90)

12. Secondary Outcome: Cognitive Control Capacity - Conflict RT Flanker
Description: The Flanker task is a psychological experiment that assesses a person's ability to focus on a target stimulus while ignoring distracting stimuli. For this measure, higher scores indicate better performance. Results reflect the difference in the reaction time between incongruent trials and congruent trials on the Flanker task.
Time Frame: Up to 4 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
Number analyzed (Participants) | 6
milliseconds | 122.58 (39.81)

13. Other Pre Specified Outcome: Feasibility/Acceptability and Experimental Outcome
Description: Outcome measures that indicate how much the video game was played and acceptability of the game as indicated by self-report ratings. Includes:
  gameplay metrics from the video game (total amount of missions completed across the 4-weeks of the intervention), Endeavor Satisfaction Survey Scores (Scale 1-5 (3 is neutral) on each item; parent and child report), and depressive symptoms at baseline (Children's Depression Inventory).
Time Frame: Up to 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Computerized Cognitive Training (CCT) Using EndeavorRx
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computerized Cognitive Training (CCT) Using EndeavorRx (N=20)
Minor neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Common cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flu (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Increase of depressive symptoms >25% on CDI from T1 to T2 (Psychiatric disorders) | 1 (1)
Increase of depression symptoms >25% on CDI from T1 to T3 (Psychiatric disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This was a small-scale study, and there was no randomization or control intervention provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT05697627/Prot_SAP_000.pdf